CLINICAL TRIAL: NCT03866265
Title: Anti-Inflammatory and Anti-Coagulant Effects of a Novel Food Grade Salmon Polar Lipids Supplement
Brief Title: Anti-Inflammatory and Anti-Coagulant Effects of Salmon Polar Lipids
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Limerick (Other)
Responsible Party: Principal Investigator, Ioannis Zabetakis, Head of the Department of Biological Sciences, University of Limerick
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Prevention
Other Study IDs: DeptBiolScULimerick
Record Dates: First submitted 2019-03-01; First posted 2019-03-07 (Actual); Last update posted 2019-12-19 (Actual); Status verified 2019-12

CONDITIONS: Platelet Thrombus
Keywords: Platelet Sensitivity; PAF; Thrombin; Salmon Polar Lipids; anti-inflammatory; anti-coagulant; platelet aggregation

STUDY DESIGN:
Intervention Model Description: Blood samples will be taken at day 0 from all Subjects. 10 of them will be administered for 28 days a food supplement capsule (0.125 g of FGE-Salmon-PLs) per day, while the other 10 will be administered a placebo capsule (0.125 g of glycerine) per day, in a double blind and randomized way.
  After 28-days, blood samples will be collected from all Subjects. No administration of any kind of capsules will follow for 14 days for all Subjects.
  After this 14-days period, blood samples will be collected from all Subjects Then, in a crossover design each participant initially on supplement will now be administered the placebo capsules, while likewise each participant initially on placebo will now be administered the supplement capsules for 28 days.
  After this new 28-days period, blood samples will be collected from all Subjects.
  All collected blood samples from each participant will be tested for their platelet sensitivity against both PAF and Thrombin induced platelet aggregation.
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Supplement Group (Active Comparator): 10 Subjects will provide baseline blood samples at day 0. Just after they will be initially administered a food supplement capsule (containing 0.125 g of FGE-Salmon-PLs) per day for a period of 28 days.
  After the period of 28 days, each participant will provide blood samples at the 29th day.
  Then a washout period of 14 days will follow, in which each participant will not be administered any kind of capsules.
  After this washout period of 14 days, each participant will provide again new baseline blood samples and then in a crossover design the participants of this group that were initially administered the food supplement will now be administered the placebo capsules for 28 days (a placebo capsule per day)
  Interventions: Dietary Supplement: Food Grade Extract of Salmon Polar Lipids (FGE-Salmon-PLs)
- Placebo Group (Placebo Comparator): 10 Subjects will provide baseline blood samples at day 0. Just after they will be initially administered a placebo capsule (containing 0.125 g of glycerin) per day for a period of 28 days.
  After the period of 28 days, each participant will provide blood samples at the 29th day.
  Then a washout period of 14 days will follow, in which each participant will not be administered any kind of capsules.
  After this washout period of 14 days, each participant will provide again new baseline blood samples and then in a crossover design the participants of this group that were initially administered the placebo capsules will now be administered the food supplement capsules for 28 days (a food supplement capsule per day)
  Interventions: Other: Placebo

INTERVENTIONS:
Dietary Supplement: Food Grade Extract of Salmon Polar Lipids (FGE-Salmon-PLs) — Each participant will be administered per day a capsule of the FGE-Salmon-PLs food supplement (containing 0.125 g of FGE-Salmon-PLs) for a period of 28 days in a double blind randomized, crossover and placebo-controlled design.
  Arms: Supplement Group
Other: Placebo — Each participant will be administered per day a placebo capsule (containing 0.125 g of glycerin) for a period of 28 days in a double blind randomized, crossover design.
  Arms: Placebo Group

SUMMARY:
Inflammation is a normal immune response to tissue healing. However, uncontrolled and unresolved inflammation can initiate and further induce several chronic manifestations that contribute to chronic disorders such as atherosclerosis and cardiovascular disease (CVD). A 'cross-talk' between platelets, endothelial cells and leukocytes, accompanied by activation and aggregation of platelets, contribute to inflammation-related atherogenic, atherosclerotic and athero-thrombotic events.

Platelet Activating Factor (PAF) and Thrombin are the most potent platelet agonists inducing platelet activation and aggregation that are also implicated in the patho-physiology of platelets and endothelium and thus in inflammation-related chronic disorders. Therefore, the inhibition of PAF and Thrombin related pathways of platelet aggregation, coagulation and inflammation provide a potential therapeutic strategy for anti-platelet, anti-coagulation and suppression of inflammatory responses in CVDs and other chronic disorders.

The investigators have previously reported bio-active lipid molecules with strong anti-PAF and anti-Thrombin effects to be present in natural, non-toxic food, microorganisms, plants and especially in several marine sources. The plethora of in vitro beneficial bio-activities of marine polar lipids (PLs) against atherosclerosis and CVDs indicate therapeutic potential. Recently, the investigators have also demonstrated that PLs extracted from Irish, organic farmed salmon (Salmo salar) display strong in vitro anti-thrombotic effects against platelet aggregation, bio-activities that were related to inhibitory effect against PAF and Thrombin pathways.

The present study investigates the putative anti-platelet effects in healthy human subjects following ingestion of a novel supplement containing food-grade extracts of bio-active salmon polar lipids (FGE-Salmon-PLs).

The study has a double blind randomized cross-over placebo-controlled design in healthy subjects.

Each Subject will be administrated the FGE-Salmon-PLs Food Supplement capsules for 28 days (a capsule containing 0.125 g of FGE-Salmon-PLs per day) and platelet sensitivity against both PAF and Thrombin will be tested in blood samples of each subject just before and after the supplement administration. The same tests will be conducted in blood samples of each participant in a crossover design before and after 28 days of placebo capsules administration (a capsule containing 0.125 g of glycerin per day).

DETAILED DESCRIPTION:
The present study investigates the putative anti-platelet effects in healthy human subjects (N=20) following ingestion of a novel supplement containing food-grade extracts of bio-active salmon polar lipids (FGE-Salmon-PLs).

The study has a double blind randomized cross-over placebo-controlled design in healthy subjects.

After appropriate screening, 20 of the recruited subjects will provide baseline blood samples and then 10 of them will be initially administered a food supplement capsule (containing 0.125 g of FGE-Salmon-PLs) per day for a period of 28 days, while another 10 of them will initially be administered a placebo capsule (containing 0.125 g of glycerin) per day, in a double blind and randomized way.

After the period of 28 days, each participant will provide blood samples at the 29th day.

Then a washout period of 14 days will follow, in which each participant will not be administered any kind of supplements or placebo capsules.

After this washout period of 14 days, each participant will provide again new baseline blood samples and then in a crossover design the participants that were initially administered the food supplement will now be administered the placebo capsules for 28 days (a placebo capsule per day), while likewise the participants that were initially administered the supplement capsules will now be administered the food supplement capsules for 28 days.

After this new period of 28 days, each participant will provide again blood samples at the new 29th day.

Plasma reach in platelets of all blood samples from each participant, before and after each kind of administration (of either placebo or supplement capsules), will be tested for their platelet sensitivity against both PAF and Thrombin induced platelet aggregation.

ELIGIBILITY:
Inclusion Criteria:

* The selection criteria of the subjects will be as follows:

  1. they need to be off medication and off intake of dietary supplements
  2. they need to have no blood clotting disorders or dyslipidaemia and

Exclusion Criteria:

Subjects with clotting disorders, dyslipidemia or being on medication (i.e. statins) or other supplements during the study will be excluded.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2019-04-01 (Actual); Primary Completion 2019-11-15 (Actual); Study Completion 2019-12-15 (Actual)

PRIMARY OUTCOMES:
Effect on the Platelet Sensitivity against PAF | Tests will be conducted just after blood collection for each blood sample and the outcomes measured will be assessed up to 6 months, for which the data will be reported through study completion
  Platelet sensitivity against PAF of platelet rich plasma of each blood sample will be determined by the % observed change of the EC50 value of PAF-induced platelet aggregation before and after administration of either the FGE-Salmon-PLs food supplement or the placebo capsules.
Effect on the Platelet Sensitivity against Thrombin | Tests will be conducted just after blood collection for each blood sample and the outcomes measured will be assessed up to 6 months, for which the data will be reported through study completion
  Platelet sensitivity against Thrombin of platelet rich plasma of each blood sample will be determined by the % observed change of the EC50 value of Thrombin-induced platelet aggregation before and after administration of either the FGE-Salmon-PLs food supplement or the placebo capsules.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Limerick, Limerick, Co. Limerick, Ireland

IPD SHARING:
Plan to Share IPD: Undecided